CLINICAL TRIAL: NCT07279246
Title: The Effects of Exercise and Music Combination on Drug Cravings, Depression and Self-Efficacy Among Drug Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WEIPENG DUAN (Other)
Responsible Party: Sponsor-Investigator, WEIPENG DUAN, Lecturer, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23010064
Record Dates: First submitted 2025-11-13; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Drug Craving Levels Among Individuals With Substance Addiction; Depression Levels Among Individuals With Substance Addiction; Self-efficacy Among Individuals With Substance Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sports group (Experimental): Participants shall engage in the standard activities required at the compulsory isolation drug rehabilitation centre, whilst researchers will supplement the subjects' regimen with an exercise therapy programme.
  Interventions: Behavioral: Sports group; Behavioral: Exercise combined with fast-paced music group; Behavioral: Exercise combined with slow-tempo music group
- Exercise combined with fast-paced music group (Experimental): Participate in the standard activities required at the compulsory isolation drug rehabilitation centre, whilst researchers will supplement the treatment regimen for subjects with exercise combined with fast-paced music.
  Interventions: Behavioral: Sports group; Behavioral: Exercise combined with fast-paced music group; Behavioral: Exercise combined with slow-tempo music group
- Exercise combined with slow-tempo music group (Experimental): Participants will engage in standard activities required at the compulsory isolation drug rehabilitation centre, whilst researchers will supplement the treatment regimen with exercise combined with slow-tempo music.
  Interventions: Behavioral: Sports group; Behavioral: Exercise combined with fast-paced music group; Behavioral: Exercise combined with slow-tempo music group

INTERVENTIONS:
Behavioral: Sports group — The intervention groups in the experiment comprised three main categories: an exercise-only group, an exercise-combined-with-fast-paced-music group, and an exercise-combined-with-slow-music group. Participants engaged in activities mandated by the compulsory isolation drug rehabilitation centre, while researchers administered three distinct treatment protocols to the subjects.
Behavioral: Exercise combined with fast-paced music group — Participate in the standard activities required at the compulsory isolation drug rehabilitation centre, whilst researchers will supplement the treatment regimen for subjects with exercise combined with fast-paced music.
Behavioral: Exercise combined with slow-tempo music group — Participants will engage in standard activities required at the compulsory isolation drug rehabilitation centre, whilst researchers will supplement the treatment regimen with exercise combined with slow-tempo music.

SUMMARY:
This study focuses on the rehabilitation of drug addicts by combining exercise and music, to find out whether exercise and exercise combined with music of different rhythms will have an improvement for drug addicts.

1. What are the Chinese translated versions of the Basic Depression Questionnaire (CBD), the Mann Craving Scale (MaCS), the Quick Inventory of Depressive Symptoms (QIDS SR-16), and the New General Self-Efficacy Scale (NGSES)?
2. Based on confirmatory factor analysis, are the Chinese versions of the CBD, MaCS, QIDS SR-16, and NGSES valid and reliable?
3. Is the concurrent validity of the translated versions of the CBD and MaCS supported when compared to the Chinese versions of the Quick Inventory of Depressive Symptoms (QIDS SR-16) and the Visual Analogue Scale (VAS), respectively?
4. Which exercise programs, fast-paced music, and slow-paced music are suitable for drug addicts?
5. is there an effect of exercise and music therapy on drug craving, depression, and self-efficacy in drug addicts (time, group, and interaction)? The researchers divided the participants into four groups: a control group; an exercise group; an exercise combined with a tempo group; and an exercise combined with a slow tempo group.

   * Scientific physical activity at a fixed time each week for 6 months
   * Conducted questionnaires and addiction level tests between each month
   * Record their emotional status and addiction level.

ELIGIBILITY:
Inclusion Criteria:

1. Drug-addicted individuals aged 18 years or older.
2. Confirmed diagnosis of drug addiction through testing and currently undergoing compulsory drug rehabilitation treatment at a compulsory isolation drug rehabilitation centre in China.
3. Educational attainment of primary school level or above and capable of independently completing questionnaires.
4. No prior occupational experience in sports or music-related fields.

Exclusion Criteria:

1. Less than six months remaining in the educational phase of compulsory isolation drug rehabilitation.
2. Presence of other severe drug addiction-related complications, such as infectious diseases (e.g., HIV/AIDS), severe cardiovascular or respiratory system diseases.
3. Presence of other conditions that may impair hearing or motor function, such as hearing impairments or medical contraindications for physical activity due to other health conditions.
4. Refusal to participate in this experimental study or refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Depression | Indicator measurements were taken from the commencement of the experiment until its conclusion, with one measurement taken prior to the experiment and subsequent monthly measurements every month thereafter, totalling seven measurements over the six-month
  Depression serves as the single core indicator under investigation, assessed via two independent scales: ① the Common Depression Questionnaire (CBD), and ② the Quick Inventory of Depressive Symptoms (QIDS-SR16).
  Both scales measure participants' depressive states, yet results will be presented and analysed separately to enhance the reliability and stability of depression symptom assessment.
  The CBD scores range from 0 to 63 points, with higher scores indicating greater severity of depression. Scores are categorised as follows: no depression (0 to 19); mild depression (20 to 29); moderate depression (30 to 39); and severe depression (40 or more).
  The QIDS-SR16 ranges from 0-27 points, with higher scores indicating greater depression severity.1-5 points: no depression; 6-10 points: mild depression;11-15 points: moderate depression; 16-20 points: severe depression; 21-27 points: very severe depression.
Drug Craving | Indicator measurements were taken from the commencement of the experiment until its conclusion, with one measurement taken prior to the experiment and subsequent monthly measurements every month thereafter, totalling seven measurements over the six-month
  This study employed the Mannheim Craving Scale (MaCS) German version and the Visual Analogue Scale (VAS) to assess participants' drug craving levels. Both instruments measure the same core indicator, "drug craving level", but were recorded and analysed as independent measurement tools to enhance measurement reliability and reflect the breadth of the dimension.
  * MaCS (German version) is a graded rating scale (scoring range: 0-48 points, with higher scores indicating stronger craving)
  * VAS visual analogue scoring employs a 0-10 cm quantitative scale, where 0 denotes complete absence of craving and 10 denotes extremely strong craving
  Measurement timepoints: One baseline measurement prior to the experiment, followed by monthly measurements during the experiment, totalling seven measurements over six months.
Self-Efficacy | Measurements were taken from the commencement of the experiment until its conclusion, with one measurement prior to the experiment and one monthly thereafter, totalling seven measurements over the six-month experimental period.
  Self-efficacy will be evaluated using the New General Self-Efficacy Scale (NGSES).
  The NGSES is a Likert-type scale with a total scores range from 8 to 40, with higher scores indicating greater perceived self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Garry Kuan, Study Chair — Universiti Sains Malaysia; weipeng duan, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Yes